CLINICAL TRIAL: NCT05420753
Title: Single-center Randomized Controlled Trial to Evaluate Body Composition Changes and Clinical Outcomes After Transjugular Intrahepatic Portosystemic Shunt (TIPS) Creation in Patients With Cirrhosis and Complications of Portal Hypertension Awaiting Liver Transplantation
Brief Title: Body Composition Changes After TIPS and Associated Clinical Outcomes
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00022853
Record Dates: First submitted 2022-05-06; First posted 2022-06-15 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cirrhosis, Liver; Sarcopenia
Keywords: cirrhosis; liver transplantation; sarcopenia; frailty
MeSH Terms: conditions — Liver Cirrhosis; Sarcopenia; Fibrosis; Frailty | interventions — Portasystemic Shunt, Transjugular Intrahepatic; Facility Design and Construction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIPS (Experimental): Patients in this arm will undergo TIPS creation in addition to their current management.
  Interventions: Procedure: Transjugular Intrahepatic Portosystemic Shunt (TIPS) creation
- Standard of care (No Intervention): Patients in this arm will continue to be treated with their current management

INTERVENTIONS:
Procedure: Transjugular Intrahepatic Portosystemic Shunt (TIPS) creation — During a TIPS procedure, the interventional radiologist, with the help of x-ray and ultrasound guidance, makes a channel through the liver to connect the portal vein (the vein that carries blood from the digestive organs to the liver) to one of the hepatic vein (three veins that carry blood away from the liver back to the heart) using a special type of needle. The interventional radiologist then replaces the needle with a wire and catheter, and a small tubular device called a stent graft is placed in this channel to keep the pathway open between the two blood vessels.
  Arms: TIPS

SUMMARY:
The purpose of this study is to prospectively assess the impact of TIPS creation on muscle mass and physical function in patients with cirrhosis, and to determine whether these changes correlate with improved outcomes in patients awaiting liver transplantation. Retrospective observational studies have shown improvement in muscle mass and body composition in cirrhotic patients undergoing TIPS. The investigators aim to now prospectively study this through a pilot randomized controlled trial tracking patients managed with TIPS creation compared to those managed without TIPS to determine whether these observational findings can be seen in a randomized cohort. The investigators hypothesize that TIPS creation will lead to improved muscle mass, body composition and muscle function within the first 12 months after the procedure compared to a control group without TIPS, and that these changes will improve liver disease outcomes in patients awaiting liver transplantation.

DETAILED DESCRIPTION:
Sarcopenia (loss of muscle mass) and frailty (loss of muscle function) have increasingly become recognized as major prognostic factors in predicting morbidity and mortality with several disease states, including cirrhosis. Cirrhosis represents end-stage liver disease and is complicated by a multitude of clinical sequelae, such as variceal hemorrhage, ascites, renal insufficiency, hepatic encephalopathy, hepatopulmonary syndrome, cardiac dysfunction, infection and hepatocellular carcinoma. To date, liver transplantation remains the only prospect for a curative treatment. As the liver is the primary metabolic organ, sarcopenia is prevalent in cirrhosis, afflicting 30-70% of patients. Observational studies have implicated sarcopenia as an independent risk factor for morbidity and mortality in all clinical sequelae of cirrhosis. Moreover, sarcopenia and frailty have been shown to increase morbidity and mortality of transplant eligible patients on the liver transplant waitlist, as well as mortality of patients after liver transplant. Given the prevalence of sarcopenia and frailty in this patient population, and the severe clinical impacts, addressing these adverse predictors may have profound implications for the outcomes of patients with cirrhosis.

Cirrhosis often leads to portal hypertension, complications of which include lower extremity edema, ascites, hepatic hydrothorax, variceal bleeding, portal hypertensive gastropathy, portal vein thrombosis, and hepatic encephalopathy. Patients with cirrhosis and complications of portal hypertension are currently managed in several ways in clinical practice:

* medical management, including diuretics and non-selective beta blocker therapy
* endoscopic options include variceal banding or glue embolization
* invasive options include large-volume paracentesis (LVP) or transjugular intrahepatic portosystemic shunt (TIPS) creation.

Since 1988, the Liver Transplant Program at OHSU has been successfully treating waitlisted cirrhotic patients with complications of portal hypertension using a combination of these therapies. TIPS creation, particularly in the current era of stent grafts with a dedicated device for this procedure, has been a part of managing patients with cirrhosis as a bridge to transplant for two decades. Depending on the indication, patients can be treated with a combination of these therapies often with significant overlap. For example, a given patient with portal hypertension and ascites may be managed with diuretics and serial LVP vs. TIPS creation, and a given patient with variceal bleeding may be treated with beta-blockers and endoscopic banding vs. TIPS creation.

Of relevance to the proposed trial, recent observational studies have demonstrated significant reversal of sarcopenia after TIPS creation, and this reversal has been strongly correlated with improved survival and less hepatic encephalopathy. Moreover, the time course of muscle gains has been observed to occur within the first 6 months of TIPS creation, critical for patients awaiting liver transplantation, as benefits would occur during typical transplant waitlist time periods. Thus, TIPS creation may represent a major unmet need to address sarcopenia and frailty in patients with cirrhosis, and represents an intervention with potential to reverse this debilitating condition and improve clinical outcomes. Putative mechanisms for how TIPS creation may improve body composition include decreased congestive enteropathy resulting in improved gut nutrient absorption, decrease in metabolic burden from a hyperdynamic cardiopulmonary status in the setting of fluid overload, improvement in renal function, and changes in the gut microbiome resulting in conversion from a catabolic to an anabolic state. A major gap in knowledge, however, remains whether TIPS creation can directly reverse muscle loss. Furthermore, whether reversal of muscle loss results in improved measures of strength, physical performance and clinical outcomes has not been prospectively studied. In this proposal, the investigators plan to address this major knowledge gap through a pilot prospective randomized controlled trial tracking patients managed with TIPS creation compared to those managed without TIPS to determine whether these observational findings can be seen in a randomized cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 <99 with cirrhosis wait listed for liver transplantation
* Evidence of complications of portal hypertension:
* Ascites or hydrothorax requiring escalation of diuretic medication
* Persistent ascites or hydrothorax despite diuretic use, or intolerance of diuretic use
* Gastrointestinal varices and blood loss anemia or history of variceal hemorrhage
* Portal hypertensive gastropathy and blood loss anemia
* Chronic portal vein thrombosis requiring recanalization and TIPS for transplant

Exclusion Criteria:

* Hepatocellular carcinoma or other active malignancy
* Recurrent overt hepatic encephalopathy
* Uncontrolled coagulopathy with maximum amplitude (MA) <30 on thromboelastography
* Bacteremia or sepsis
* MELD > 25
* Pregnant
* Decisionally impaired individuals
* Need for emergency TIPS creation
* Patients who do not have acceptable alternatives to TIPS creation to manage their disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Body composition changes | Start to 2 years after enrollment
  Muscle and fat content as assessed by CT scan
Short Performance Physical Battery test | Start to 6 months after enrollment
  Brief physical test for balance with feet together (seconds), gait speed walking 4 meters (seconds), time to stand from a chair (seconds). These are aggregated together to a unified score.
Liver Frailty test | Start to 6 months after enrollment
  Brief physical test for balance with feet together (seconds), time to stand from a chair (seconds), and grip strength (kilograms of force). These are aggregated together to a unified score.

SECONDARY OUTCOMES:
Chronic Liver Disease Quality of Life Questionnaire | Start to 6 months after enrollment
  Quality of life assessment using 29 questions regarding experience of various symptoms graded on a scale of 1-7 each, with 1 being worse (all of the time) and 7 being the best (none of the time).
Overall survival | Start to 2 years after enrollment
  Survival time
Transplant complications | Start to 30 days after transplant
  Complications while on transplant waitlist as well as after transplant
Cardiac function | Start to 6 months after enrollment
  Right and left ventricular function noted by echocardiography
Liver function tests | Start to 6 months after enrollment
  Serum tests for total bilirubin (mg/dL), albumin (g/dL), sodium (mmol/L), creatinine (mg/dL), international normalized ratio. These values will be combined in the MELD score = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43, and MELD-Na score = MELD + 1.32 x (137 - Na) - [0.033 x MELD*(137 - Na)]
Cardiac mass | start to 6 months after enrollment
  Myocardial mass as measured by echocardiography
Serum ammonia | start to 6 months after enrollment
  serum ammonia level (micromol/L)
Serum glucose | start to 6 months after enrollment
  serum glucose level (mg/dL)

OTHER OUTCOMES:
Stool microbiome genomic assessment | Start to 6 months after enrollment
  Stool sample using DNAGenotek Omni-gene Stool collection kit to assess for bacterial complement in stool
Lipocalin-2 biomarker assessment | Start to 6 months after enrollment
  Lipocalin-2 transcription and expression (RNA sequencing/Elisa/Western Blot) in serum samples
IL-6 biomarker assessment | Start to 6 months after enrollment
  IL-6 immunoassay assessment of serum (pg/mL)
Salivary cortisol biomarker assessment | Start to 6 months after enrollment
  salivary cortisol (mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States